CLINICAL TRIAL: NCT04914039
Title: Evaluation of CTA on the Assessment of Brain Death
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-031
Record Dates: First submitted 2021-06-01; First posted 2021-06-04 (Actual); Last update posted 2021-06-04 (Actual); Status verified 2021-05

CONDITIONS: Brain Death
Keywords: brain death; CT angiography
MeSH Terms: conditions — Brain Death | interventions — Piperacillin, Tazobactam Drug Combination

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- CTA examination: CTA examination group for suspected brain death
  Interventions: Combination Product: Combination Product
- Confirmed: Confirmed group for brain death
  Interventions: Other: NO CTA examination

INTERVENTIONS:
Combination Product: Combination Product — Cases of brain death confirmed by the classic brain death confirmation test
  Groups: CTA examination
Other: NO CTA examination — NO CTA examination
  Groups: Confirmed

SUMMARY:
At present, different countries have different standards for the diagnosis of brain death, but according to the classic brain death confirmation test, it needs to be combined with transcranial Doppler, EEG, evoked potential and apnea test in clinical practice. Some patients cannot undergo a complete clinical examination and apnea test due to certain factors, and the determination of brain death is limited. The American Academy of Neurology (AAN) guidelines regard cerebral angiography as an acceptable auxiliary examination and is widely regarded as the gold standard for cerebral blood flow evaluation. CT cerebrovascular angiography (CTA) is a noninvasive and widely used examination method that can identify missing or severely reduced cerebral blood flow. However, due to limited experience and lack of sufficient evidence to prove its reliability, it is not included in the AAN A recognized auxiliary examination; there are also a large number of domestic and foreign literature reports that CTA can be used as a new confirmation test for clinical judgment of brain death.

This study aims to explore the value of CTA in the judgment of patients with brain death.

ELIGIBILITY:
Inclusion Criteria:

* Recruiting, no definite

Exclusion Criteria:

* Recruiting, no definite

Ages: 12 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: CTA imaging data of 63 patients with clinically suspected brain death
Sampling Method: Probability Sample
Enrollment: 63 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-02-01 (Estimated); Study Completion 2023-02-01 (Estimated)

PRIMARY OUTCOMES:
CTA used as an auxiliary diagnosis to determine brain death | through study completion, an average of 3 years.
  CTA used as an auxiliary diagnosis to determine brain death

CONTACTS AND LOCATIONS:
Locations (1):
- Brain Center, Second Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided